CLINICAL TRIAL: NCT06424639
Title: A Randomized, Controlled Trial Comparing the Safety and Efficacy of Luspatercept Plus Cyclosporine Versus Cyclosporine Alone for the Treatment of Newly Diagnosed Non-transfusion-dependent Non-severe Aplastic Anemia (NSAA)
Brief Title: Luspatercept Plus CsA vs CsA for the Treatment of Newly Diagnosed Non-Transfusion-Dependent NSAA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC-001
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia; Luspatercept; CsA; randomized controlled study
MeSH Terms: conditions — Anemia, Aplastic | interventions — luspatercept; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Luspatercept combined with cyclosporine (Experimental): Administered Luspatercept (1.0 mg/kg, subcutaneous injection every 3 weeks), and Cyclosporine (3-5mg/kg/day) adjusted according to hematological parameters, for at least 6 months to evaluate efficacy. Effective patients will continue to receive Cyclosporine treatment for at least 1.5 years, followed by a gradual reduction in dosage.
  Interventions: Drug: Luspatercept; Drug: cyclosporine
- cyclosporine (Experimental): Give cyclosporine 3-5mg/kg/day, adjust the dose based on the blood count, and administer it for at least 6 months to evaluate the efficacy. If effective, the patient will continue to receive cyclosporine treatment for at least 1.5 years, followed by a gradual reduction in dosage.
  Interventions: Drug: cyclosporine

INTERVENTIONS:
Drug: Luspatercept — Luspatercept (dose of 1.0 mg/kg, subcutaneous injection every 3 weeks) Cyclosporine (3-5mg/kg/day)
  Other Names: cyclosporine
  Arms: Luspatercept combined with cyclosporine
Drug: cyclosporine — Cyclosporine (3-5mg/kg/day)

SUMMARY:
In a randomized, controlled clinical trial, the efficacy and safety of rodsipil combined with cyclosporine versus cyclosporine alone in the treatment of newly diagnosed non-transfusion-dependent NSAA were compared.

DETAILED DESCRIPTION:
Conduct a comparative evaluation of the effectiveness and safety of Luspatercept combined with cyclosporine versus cyclosporine monotherapy in the treatment of newly diagnosed non-transfusion-dependent non-severe aplastic anemia (NSAA). Patients were randomized in a 1:1 ratio and assigned to one of two groups: Group A, Luspatercept combined with cyclosporine: received Luspatercept (1.0 mg/kg, subcutaneous injection every 3 weeks), cyclosporine (3-5mg/kg/day), adjusted based on hematological parameters, for at least 6 months to assess efficacy. Effective patients continued to receive cyclosporine treatment for at least 1.5 years, with a gradual reduction in dosage; Group B, cyclosporine: received 3-5mg/kg/day, adjusted based on hematological parameters, for at least 6 months to assess efficacy, with effective patients continuing to receive cyclosporine treatment for at least 1.5 years, with a gradual reduction in dosage. Hgb below 60g/L was allowed, or in emergency conditions, blood transfusion was allowed. Platelets below 20×10^9/L or with obvious bleeding tendency were allowed to receive platelet transfusion. If neutrophil count was below 1.0×10^9/L, G-CSF was allowed until neutrophil count recovered to above 1.0×10^9/L. Symptoms, treatment-related adverse events, signs, blood transfusion volume, and laboratory tests (including reticulocyte count) were recorded at least every 3 months for the first 3 months, and every 6 months thereafter until 6 months, and bone marrow aspiration, biopsy, and chromosome examination were performed at least every 6 months to observe efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Hemoglobin level of 6-10 g/dL
3. Definition of NSAA: Patients with AA diagnosis but not SAA or VSAA diagnosis (at least two of the following conditions can be diagnosed as AA: (i) Hemoglobin < 100 g/L; (ii) Platelet count < 50×10^9/L; (iii) Neutrophil count < 1.5×10^9/L. SAA diagnosis criteria include less than 25% (or 25-50%, but residual hematopoietic cells < 30%) of bone marrow cells, plus at least two of the following conditions: (i) Neutrophil count < 0.5×10^9/L; (ii) Platelet count < 20×10^9/L; (iii) Retroperitoneal lymph node count < 20×10^9/L. VSAA meets the criteria for SAA, but with neutrophil count < 0.2×10^9/L. (British guidelines, 2015))
4. No active infection
5. No other concurrent neoplasms (except in situ carcinoma)
6. Baseline liver and renal function within 1.5 times of normal value
7. No pregnancy or breastfeeding
8. Agree to sign informed consent form
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

1. Congenital aplastic anemia
2. Presence of chromosomal aberrations
3. Cytogenetic evidence of clonal hematological myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML)
4. PNH clone ≥50%
5. Previous use of alemtuzumab, any ATG, or any dose of cyclosporine for immunosuppressive treatment
6. Previous hematopoietic stem cell transplant (HSCT)
7. Uncontrolled infection or bleeding under standard treatment
8. Allergy to rituximab, cyclosporine, or excipients
9. History of allergy to polyethylene glycol (PEG) 80
10. Active infection or cirrhosis of the liver or portal hypertension due to HIV, HCV, or HBV
11. Screening QTcF (Fridericia QT corrected formula) less than 450 milliseconds or less than 480 milliseconds of bundle branch block determined by three ECG averages, and assessed on-site; unstable angina; uncontrolled hypertension (>180/100 mmHg); pulmonary hypertension
12. Any malignant tumor within 5 years, except local basal cell carcinoma; previous thromboembolic event, history of myocardial infarction or stroke (including antiphospholipid syndrome); currently using anticoagulants
13. Pregnant or lactating women
14. Participated in another clinical trial within 3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | 6 month
  Proportion of patients who achieved complete response, partial response and hematological response

SECONDARY OUTCOMES:
overall response rate (ORR) | 12 month
  Proportion of patients who achieved complete response, partial response and hematological response
adverse event rate | 12 month
  Proportion of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bing Bing, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young NS. Aplastic anaemia. Lancet. 1995 Jul 22;346(8969):228-32. doi: 10.1016/s0140-6736(95)91273-8. No abstract available. PMID 7616805
- [Background] Young NS. Aplastic Anemia. N Engl J Med. 2018 Oct 25;379(17):1643-1656. doi: 10.1056/NEJMra1413485. No abstract available. PMID 30354958
- [Background] Bacigalupo A. How I treat acquired aplastic anemia. Blood. 2017 Mar 16;129(11):1428-1436. doi: 10.1182/blood-2016-08-693481. Epub 2017 Jan 17. PMID 28096088
- [Background] Yang C, Zhang X. Incidence survey of aplastic anemia in China. Chin Med Sci J. 1991 Dec;6(4):203-7. PMID 1813058
- [Background] Vaht K, Goransson M, Carlson K, Isaksson C, Lenhoff S, Sandstedt A, Uggla B, Winiarski J, Ljungman P, Brune M, Andersson PO. Incidence and outcome of acquired aplastic anemia: real-world data from patients diagnosed in Sweden from 2000-2011. Haematologica. 2017 Oct;102(10):1683-1690. doi: 10.3324/haematol.2017.169862. Epub 2017 Jul 27. PMID 28751565
- [Background] Li H, Fu L, Yang B, Chen H, Ma J, Wu R. Cyclosporine Monotherapy in Pediatric Patients With Non-severe Aplastic Anemia: A Retrospective Analysis. Front Med (Lausanne). 2022 Mar 7;9:805197. doi: 10.3389/fmed.2022.805197. eCollection 2022. PMID 35342744
- [Background] Kubasch AS, Fenaux P, Platzbecker U. Development of luspatercept to treat ineffective erythropoiesis. Blood Adv. 2021 Mar 9;5(5):1565-1575. doi: 10.1182/bloodadvances.2020002177. PMID 33687432
- [Background] Attie KM, Allison MJ, McClure T, Boyd IE, Wilson DM, Pearsall AE, Sherman ML. A phase 1 study of ACE-536, a regulator of erythroid differentiation, in healthy volunteers. Am J Hematol. 2014 Jul;89(7):766-70. doi: 10.1002/ajh.23732. Epub 2014 Apr 26. PMID 24715706
- [Background] Suragani RN, Cadena SM, Cawley SM, Sako D, Mitchell D, Li R, Davies MV, Alexander MJ, Devine M, Loveday KS, Underwood KW, Grinberg AV, Quisel JD, Chopra R, Pearsall RS, Seehra J, Kumar R. Transforming growth factor-beta superfamily ligand trap ACE-536 corrects anemia by promoting late-stage erythropoiesis. Nat Med. 2014 Apr;20(4):408-14. doi: 10.1038/nm.3512. Epub 2014 Mar 23. PMID 24658078
- [Background] Markham A. Luspatercept: First Approval. Drugs. 2020 Jan;80(1):85-90. doi: 10.1007/s40265-019-01251-5. PMID 31939073
- [Background] Fenaux P, Platzbecker U, Mufti GJ, Garcia-Manero G, Buckstein R, Santini V, Diez-Campelo M, Finelli C, Cazzola M, Ilhan O, Sekeres MA, Falantes JF, Arrizabalaga B, Salvi F, Giai V, Vyas P, Bowen D, Selleslag D, DeZern AE, Jurcic JG, Germing U, Gotze KS, Quesnel B, Beyne-Rauzy O, Cluzeau T, Voso MT, Mazure D, Vellenga E, Greenberg PL, Hellstrom-Lindberg E, Zeidan AM, Ades L, Verma A, Savona MR, Laadem A, Benzohra A, Zhang J, Rampersad A, Dunshee DR, Linde PG, Sherman ML, Komrokji RS, List AF. Luspatercept in Patients with Lower-Risk Myelodysplastic Syndromes. N Engl J Med. 2020 Jan 9;382(2):140-151. doi: 10.1056/NEJMoa1908892. PMID 31914241
- [Background] Feld J, Navada SC, Silverman LR. Myelo-deception: Luspatercept & TGF-Beta ligand traps in myeloid diseases & anemia. Leuk Res. 2020 Oct;97:106430. doi: 10.1016/j.leukres.2020.106430. Epub 2020 Jul 30. PMID 32763582
- [Background] Komrokji RS, Platzbecker U, Fenaux P, Zeidan AM, Garcia-Manero G, Mufti GJ, Santini V, Diez-Campelo M, Finelli C, Jurcic JG, Greenberg PL, Sekeres MA, DeZern AE, Savona MR, Shetty JK, Ito R, Zhang G, Ha X, Backstrom JT, Verma A. Luspatercept for myelodysplastic syndromes/myeloproliferative neoplasm with ring sideroblasts and thrombocytosis. Leukemia. 2022 May;36(5):1432-1435. doi: 10.1038/s41375-022-01521-4. Epub 2022 Feb 26. No abstract available. PMID 35220402
- [Background] Hellstrom-Lindberg E, Gulbrandsen N, Lindberg G, Ahlgren T, Dahl IM, Dybedal I, Grimfors G, Hesse-Sundin E, Hjorth M, Kanter-Lewensohn L, Linder O, Luthman M, Lofvenberg E, Oberg G, Porwit-MacDonald A, Radlund A, Samuelsson J, Tangen JM, Winquist I, Wisloff F; Scandinavian MDS Group. A validated decision model for treating the anaemia of myelodysplastic syndromes with erythropoietin + granulocyte colony-stimulating factor: significant effects on quality of life. Br J Haematol. 2003 Mar;120(6):1037-46. doi: 10.1046/j.1365-2141.2003.04153.x. PMID 12648074